CLINICAL TRIAL: NCT03101579
Title: Intrathecal Pemetrexed for Recurrent Leptomeningeal Metastasis From Non-small Cell Lung Cancer: A Prospective Pilot Clinical Trial
Brief Title: Intrathecal Pemetrexed for Recurrent Leptomeningeal Metastases From Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPRLM
Record Dates: First submitted 2017-03-23; First posted 2017-04-05 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Leptomeningeal Metastases
Keywords: Leptomeningeal metastasis; Recurrence; Intrathecal chemotherapy; Pemetrexed
MeSH Terms: conditions — Meningeal Carcinomatosis; Recurrence | interventions — Pemetrexed; Dexamethasone; Folic Acid; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-pemetrexed (Experimental): Patients were treated with intrathecal pemetrexed at dose escalation. The regimen of intrathecal pemetrexed is 10/15/20 mg, plus dexamethasone 5 mg, twice per week for 2 weeks, followed by once per week for 2-4 weeks. Pemetrexed is administrated by intrathecal injection via lumbar puncture. Folic acid 200-400 μg is administered orally once daily, prior to the first intrathecal pemetrexed, until 21 days after the last intrathecal pemetrexed. A single dose of vitamin B12 1000 μg is administered by intramuscular injection before the first intrathecal pemetrexed，once per 3 weeks. To detect the pharmacokinetics of intrathecal pemetrexed, the serum and cerebrospinal fluid samples are collected. These samples would be analyzed by spectrometer for drug concentration.
  Interventions: Drug: Pemetrexed; Drug: Dexamethasone; Drug: Folic Acid; Drug: Vitamin B12

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed,10-15 mg, intrathecal injection via lumbar puncture, twice per week for 2 weeks, followed by once per week for 2-4 weeks.
Drug: Dexamethasone — Dexamethasone, 5 mg, intrathecal injection via lumbar puncture, simultaneously with pemetrexed, twice per week for 2 weeks, followed by once per week for 2-4 weeks.
Drug: Folic Acid — Folic acid, 400 μg, oral, once per day, prior to the first intrathecal pemetrexed, until 21 days after the last intrathecal pemetrexed.
Drug: Vitamin B12 — A single dose of vitamin B12 1000 μg, intramuscular injection, before the first intrathecal pemetrexed.

SUMMARY:
It has been proved that intrathecal chemotherapy is the main treatment strategy for leptomeningeal metastases. At present, the commonly used drugs for intrathecal chemotherapy include methotrexate, cytarabine, and liposomal cytarabine. In recent decades, no new effective drugs have been discovered for intrathecal chemotherapy. The recurrence of leptomeningeal metastases is inevitable even after aggressive treatment. There is no effective treatment for recurrent leptomeningeal metastases after comprehensive treatment which includes intrathecal methotrexate and/or cytarabine, central nervous system radiation therapy, systemic chemotherapy as well as tyrosine-kinase inhibitor drugs. The quality of life is extremely poor, and the patients always die in short time. Pemetrexed is a newer multitargeted antifolate which has shown activity in various tumors. It has higher effectiveness and safety, which has been used as the first-line treatment of non-small cell lung cancer. In animal studies, pemetrexed was demonstrated to suppress tumor growth completely in mice with two types of transplanted human colon xenografts resistant to methotrexate. Therefore, the purpose of the study is to evaluate the safety and feasibility of intrathecal pemetrexed in patients with recurrent leptomeningeal metastases from non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a single arm clinical trial. The objective of the study is patients with recurrent or progressive leptomeningeal metastases from non-small cell lung cancer after leptomeningeal metastases-related treatment. The regimen of pemetrexed (Alimta, Eli Lilly and Company) is 10/15/20 mg, plus dexamethasone 5 mg, twice per week for 2 weeks, followed by once per week for 2-4 weeks. Pemetrexed and dexamethasone are administrated by intrathecal injection via lumbar puncture. Folic acid and vitamin B12 are administered to reduce the frequency of myelosuppression. Folic acid 200-400 μg is administered orally once daily, prior to the first intrathecal pemetrexed, until 21 days after the last intrathecal pemetrexed. A single dose of vitamin B12 1000 μg is administered by intramuscular injection before the first intrathecal pemetrexed，once per 3 weeks. To detect the pharmacokinetics of intrathecal pemetrexed, the serum and cerebrospinal fluid samples are collected. These samples would be analyzed by spectrometer for drug concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as leptomeningeal metastases from non-small cell lung cancer had been received comprehensive treatment, including intrathecal methotrexate and/or cytarabine, central nervous system radiation therapy, systemic chemotherapy as well as tyrosine-kinase inhibitor drugs.
2. Patients diagnosed with recurrent leptomeningeal metastases by positive cerebrospinal fluid cytological examination and persist aggravate symptoms for more than 1 week, or increased intracranial pressure (>300 mmH2O).
3. No severe abnormal liver and kidney function; WBC≥2500/mm3, Plt≥60000/mm3;
4. No other severe chronic diseases;
5. No severe dyscrasia.
6. Signed informed consent form.

Exclusion Criteria:

1. Patients with the clinical manifestation of nervous system failure including severe encephalopathy, grade III-IV white matter lesions confirmed by imaging examination, moderate or severe coma, and glasgow coma score less than 9 points;
2. Patients with severe nervous system injury related with treatment, such as chemical meningitis;
3. Patients who had accepted systemic chemotherapy within two weeks, or new molecular targeted therapeutic drug less than one months;
4. Patients with poor compliance, or for other reasons, the researchers considered unsuitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2019-01-05 (Actual)

PRIMARY OUTCOMES:
Incidence of severe adverse events | Two months after the treatment.
  Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE, version 3.0). Events of grade 3-5 are defined as moderate and severe adverse events.
Maximal tolerated dose | From the beginning of the treatment until two months after the treatment.
  A dose-limiting toxicity (DLT) was defined as grade 3 neurological toxicities (e.g. chemical meningitis) or other grade 4 toxicity. If more than two patients experienced a DLT, that level was considered too toxic. The maximal tolerated dose (MTD) was exceeded and an additional three patients should be treated at the next lower dose level. The MTD was defined as the dose where 0/3 or 1/6 patients experienced a DLT with at least two patients encountering DLT at the higher dose.

SECONDARY OUTCOMES:
Clinical response rate | One month after the treatment.
  The RANO proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Pan, Professor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Result] McDonald AC, Vasey PA, Adams L, Walling J, Woodworth JR, Abrahams T, McCarthy S, Bailey NP, Siddiqui N, Lind MJ, Calvert AH, Twelves CJ, Cassidy J, Kaye SB. A phase I and pharmacokinetic study of LY231514, the multitargeted antifolate. Clin Cancer Res. 1998 Mar;4(3):605-10. PMID 9533527
- [Result] Taylor EC, Kuhnt D, Shih C, Rinzel SM, Grindey GB, Barredo J, Jannatipour M, Moran RG. A dideazatetrahydrofolate analogue lacking a chiral center at C-6, N-[4-[2-(2-amino-3,4-dihydro-4-oxo-7H-pyrrolo[2,3-d]pyrimidin-5- yl)ethyl]benzoyl]-L-glutamic acid, is an inhibitor of thymidylate synthase. J Med Chem. 1992 Nov 13;35(23):4450-4. doi: 10.1021/jm00101a023. PMID 1447744
- [Result] Adjei AA. Pharmacology and mechanism of action of pemetrexed. Clin Lung Cancer. 2004 Apr;5 Suppl 2:S51-5. doi: 10.3816/clc.2004.s.003. PMID 15117425
- [Result] Rinaldi DA, Burris HA, Dorr FA, Woodworth JR, Kuhn JG, Eckardt JR, Rodriguez G, Corso SW, Fields SM, Langley C, et al. Initial phase I evaluation of the novel thymidylate synthase inhibitor, LY231514, using the modified continual reassessment method for dose escalation. J Clin Oncol. 1995 Nov;13(11):2842-50. doi: 10.1200/JCO.1995.13.11.2842. PMID 7595747
- [Result] Yan J, Zhong N, Liu G, Chen K, Liu X, Su L, Singhal S. Usp9x- and Noxa-mediated Mcl-1 downregulation contributes to pemetrexed-induced apoptosis in human non-small-cell lung cancer cells. Cell Death Dis. 2014 Jul 3;5(7):e1316. doi: 10.1038/cddis.2014.281. PMID 24991768
- [Result] Ramirez JM, Ocio EM, San Miguel JF, Pandiella A. Pemetrexed acts as an antimyeloma agent by provoking cell cycle blockade and apoptosis. Leukemia. 2007 Apr;21(4):797-804. doi: 10.1038/sj.leu.2404599. Epub 2007 Feb 22. PMID 17315026
- [Result] Pan Z, Yang G, He H, Zhao G, Yuan T, Li Y, Shi W, Gao P, Dong L, Li Y. Concurrent radiotherapy and intrathecal methotrexate for treating leptomeningeal metastasis from solid tumors with adverse prognostic factors: A prospective and single-arm study. Int J Cancer. 2016 Oct 15;139(8):1864-72. doi: 10.1002/ijc.30214. Epub 2016 Jun 30. PMID 27243238
- [Derived] Pan Z, Yang G, Cui J, Li W, Li Y, Gao P, Jiang T, Sun Y, Dong L, Song Y, Zhao G. A Pilot Phase 1 Study of Intrathecal Pemetrexed for Refractory Leptomeningeal Metastases From Non-small-cell Lung Cancer. Front Oncol. 2019 Aug 30;9:838. doi: 10.3389/fonc.2019.00838. eCollection 2019. PMID 31544065